CLINICAL TRIAL: NCT03266133
Title: Sleep Intervention to Improve Glycemic Control in Women With Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Roxanna Twedt, Graduate Medical Fellow, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO17050233
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Gestational Diabetes Mellitus; Sleep education
MeSH Terms: conditions — Diabetes, Gestational | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Education Intervention (Experimental): This is a two-session program designed to educate patients about healthy sleep in respect to timing, regularity, efficiency, and duration in order to promote sleep during pregnancy.
  Interventions: Behavioral: Sleep Education for Pregnancy
- Routine Care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Sleep Education for Pregnancy — Sleep education specific to pregnancy
  Arms: Sleep Education Intervention

SUMMARY:
This is a pilot randomized controlled trial involving a sleep education intervention in women with gestational diabetes to study whether sleep education during pregnancy leads to improvement in glycemic control in women with gestational diabetes and improvement in sleep duration.

DETAILED DESCRIPTION:
Patients will be identified from the Maternal-Fetal Medicine office and the Perinatal Assessment Clinic at Magee-Womens Hospital, University of Pittsburgh Medical Center. Patients with gestational diabetes will be recruited following general education regarding gestational diabetes in pregnancy which is universally done for all patients at the time of their diagnosis of gestational diabetes. Eligible subjects will be randomized to two groups (usual care vs. sleep education program).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female
2. Ages 18-50
3. Gestational age between 16 0/7 weeks and 31 6/7 weeks
4. New diagnosis of GDM, not on treatment (i.e., insulin, glyburide, or metformin) at the time of enrollment

Exclusion Criteria:

1. Children less than 18 years of age
2. Non-English speaking
3. Multiple gestations (twins, triplets, etc)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 3-6 months during pregnancy
  Proportion of participants achieving glycemic control at study end. Glycemic control defined as greater than 75% of weeks with average fasting blood glucose < 95 mg/dL and 1-hr postprandial blood glucose <140 mg/dL.
Self-reported sleep duration | 3-6 months during pregnancy
  Proportion of patients who report sleeping between 7-9 hours per night

SECONDARY OUTCOMES:
Average fasting glucose values | 3-6 months during pregnancy
Average postprandial glucose values | 3-6 months during pregnancy
Gestational age at delivery | Time of delivery
Neonatal birth weight | Time of delivery
Indication for delivery | Time of delivery
  Medical records will be used to determine whether a patient when into spontaneous labor, had an induction or labor or a recommended delivery by cesarean section. If the patient had an induction or labor or a recommended cesarean delivery, the indication for this recommendation will be recorded.
Route of delivery | Time of delivery
  Medical records will be reviewed to determine if the patient had a vaginal delivery or cesarean delivery.
Preeclampsia | Time of delivery
  Medical records will be reviewed to determine whether a patient had a diagnosis of preeclampsia prior to delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Roxanna Twedt, MD, Principal Investigator — Clinical Fellow, Division of Maternal-Fetal Medicine
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Facco FL, Parker CB, Reddy UM, Silver RM, Koch MA, Louis JM, Basner RC, Chung JH, Nhan-Chang CL, Pien GW, Redline S, Grobman WA, Wing DA, Simhan HN, Haas DM, Mercer BM, Parry S, Mobley D, Hunter S, Saade GR, Schubert FP, Zee PC. Association Between Sleep-Disordered Breathing and Hypertensive Disorders of Pregnancy and Gestational Diabetes Mellitus. Obstet Gynecol. 2017 Jan;129(1):31-41. doi: 10.1097/AOG.0000000000001805. PMID 27926645
- [Background] Twedt R, Bradley M, Deiseroth D, Althouse A, Facco F. Sleep Duration and Blood Glucose Control in Women With Gestational Diabetes Mellitus. Obstet Gynecol. 2015 Aug;126(2):326-331. doi: 10.1097/AOG.0000000000000959. PMID 26241422
- [Background] Facco FL, Grobman WA, Kramer J, Ho KH, Zee PC. Self-reported short sleep duration and frequent snoring in pregnancy: impact on glucose metabolism. Am J Obstet Gynecol. 2010 Aug;203(2):142.e1-5. doi: 10.1016/j.ajog.2010.03.041. Epub 2010 May 26. PMID 20510182
- [Background] Qiu C, Enquobahrie D, Frederick IO, Abetew D, Williams MA. Glucose intolerance and gestational diabetes risk in relation to sleep duration and snoring during pregnancy: a pilot study. BMC Womens Health. 2010 May 14;10:17. doi: 10.1186/1472-6874-10-17. PMID 20470416